CLINICAL TRIAL: NCT02825160
Title: Drug Use Investigation of Ventavis for Pulmonary Arterial Hypertension (PAH)
Brief Title: Non-interventional, Postauthorization Safety Study of Ventavis for Pulmonary Arterial Hypertension (PAH)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17941
Record Dates: First submitted 2016-06-15; First posted 2016-07-07 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Hypertension, Pulmonary
Keywords: Iloprost; Ventavis; Prostacycline analogue; Pulmonary arterial hypertension; Japan; Post-marketing surveillance
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Iloprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ventavis: Ventavis treatment group
  Interventions: Drug: Ventavis (Iloprost, BAYQ6256)

INTERVENTIONS:
Drug: Ventavis (Iloprost, BAYQ6256) — The treatment of Ventavis should comply with the local product information

SUMMARY:
This study is collecting post-marketing information on the safety and effectiveness of Ventavis under the routine clinical practice for patients with PAH

DETAILED DESCRIPTION:
This local, prospective, non-interventional, company sponsored, multi-center, single-cohort study includes patients treated with Ventavis for PAH. A total of 270 patients (valid for safety analysis) is planned to be enrolled in 5 years. Target population is patients with PAH diagnosis. This study is performed as an all-patient investigation, therefore all patients who receive Ventavis treatment for PAH need to be registered. The treatment should be performed based on the product label in Japan. The standard observation period will last for 12 months from starting Ventavis treatment. In addition, the extension observation will be carried out as long as Ventavis treatment continues or at most for more 4 years. The standard observation points are 3 month and

1 to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PAH
* Patients for whom the decision to initiate treatment with Ventavis was made as per investigator's routine treatment practice.

Exclusion Criteria:

- N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population includes PAH patients treated with Ventavis. This study is performed as an all-case investigation. Therefore, all patients who have been treated with Ventavis for PAH need to be registered in principle, until the target number of patients reached.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAE) of special interest. | Up to 5 years
  TEAE of special interest:
  * Hypotension
  * Syncope
  * Local irritation
  * Bleeding events
  * Thrombocytopenia
  * Tachycardia
Number of participants with adverse drug reaction | Up to 5 years

SECONDARY OUTCOMES:
Change from baseline in Pulmonary Vascular Resistance (PVR) after 3 and 12 months | Baseline and 3 months,Baseline and 12 months,
Change from baseline in 6-Minute Walking Distance after 3 and 12 months | Baseline and 3 months,Baseline and 12 months
Change from baseline in tricuspid regurgitation pressure gradient (TRPG) after 3 and 12 months | Baseline and 3 months,Baseline and 12 months
Change in blood concentration from baseline in brain natriuretic peptide / N-terminal pro-brain natriuretic peptide (BPN/NT-pro BNP) after 3 and 12 months. | Baseline and 3 months,Baseline and 12 months
Change from baseline in WHO functional class after 3 and 12 months | Baseline and 3 months,Baseline and 12 months,
Time to Clinical Worsening | Up to 5 years
  The 1st occurrence date of one of the following events is recorded and used for the calculation of time to clinical worsening:
  * Death (all-cause mortality), -Heart/lung transplantation, -Atrial Septostomy,
  * Hospitalization due to persistent worsening of Pulmonary Hypertension (PH),
  * Start of new PH specific treatment or modification of a preexisting Prostacycline analogues treatment except Ventavis due to worsening PH,
  * Persistent decrease in 6MWD due to worsening PH,
  * Persistent worsening of WHO functional class due to deterioration of PH

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.